CLINICAL TRIAL: NCT01641588
Title: Are You Sitting Down: Cognitive Exectutive Function Task Comparison Between Seated and Standing Positions Using Assessments From CNS Vital Signs Test Battery
Brief Title: Are You Sitting Down: Cognitive Exectutive Function Task Comparison Between Seated and Standing Positions
Acronym: sitstandcef
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Southampton (Other)
Collaborators: Royal Academy of Engineering (Unknown); Microsoft Research (Industry)
Responsible Party: Principal Investigator, M C Schraefel, Professor, University of Southampton
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1497; RAEngSRF (Other Grant/Funding Number: Royal Academy of Engineering & Microsoft Research)
Record Dates: First submitted 2012-07-11; First posted 2012-07-17 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: (Focus) Posture Effect on Cognitive Performance
Keywords: cognitive executive function; posture; cognitive performance; heart rate; eeg
MeSH Terms: interventions — Standing Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: posture: sitting or standing — Intervention: postural position - whether seated or standing. The person carries out a battery of cognitive executive functioning assessments delivered via a laptop and carried out with the laptop keyboard while either seated or standing.
  Other Names: (no other names)

SUMMARY:
The aim of this trial has been to explore the effects of self-positioning on cognitive performance in the work environment using a standardized cognitive test battery to evaluate executive function under two conditions: sitting and standing.

DETAILED DESCRIPTION:
The aim of this trial has been to explore the effects of self-positioning on cognitive performance in the work environment using a standardized cognitive test battery to evaluate executive function under two conditions: sitting and standing.

Methods: This counterbalanced controlled trial involved 17 men (mean age +/-SD: 29.8 +/- 5.5) all with a science background and graduate degrees. The participants were accustomed to working in an open environment and none of whom currently using standing desks. We used a modified version of the CNS Vital Signs (CNSVS) test battery to assess cognitive executive function (CEF) in two typical work positions - standing and seated. Participants were randomly assigned to a standing or seated position to begin the testing procedure. Upon completion of the first test round they were instructed to rest for 10 min. in a dark room with no distractions before commencing the second round of testing positioned in the alternate fashion. The main outcome measure was a CNSVS score in each of the six CEF domains in the two different work positions

ELIGIBILITY:
Inclusion Criteria:

* male
* computer savvy
* advanced education degree

Exclusion Criteria:

* ADD
* on any medication
* currently a person who uses a standing desk

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2012-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
evidence of postural effect on cognitive performance | within the hour
  use of standard cognitive exectutive function measures carried out in seated / standing position.

SECONDARY OUTCOMES:
Interaction between posture and phyiological state against cognitive executive function performance | with the hour
  Other key measures that will be used to evaluate the intervention are heart rate variablility, heart rate and eeg.

CONTACTS AND LOCATIONS:
Overall Officials: m.c. schraefel, phd, Principal Investigator — University of Southampton
Locations (1):
- University of Southampton, Southampton, Hampshire, United Kingdom

REFERENCES:
- See also: initial tech report related to this study — http://eprints.soton.ac.uk/340535/